CLINICAL TRIAL: NCT02824094
Title: Crizotinib (Xalkori (Registered)) Expanded Access Protocol For The Treatment Of Japanese Patients With Advanced Non-small Cell Lung Cancer (Nsclc) Harboring A Translocation Or Inversion Involving The Ros1 Oncogene
Brief Title: Crizotinib Expanded Access Protocol For ROS1 Positive NSCLC
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8081064
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Expanded Access Protocol; crizotinib; Xalkori; ROS1; Japanese; A8081064
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

INTERVENTIONS:
Drug: crizotinib — Crizotinib, 250 mg BID, will be administered orally on a continuous daily dosing schedule

SUMMARY:
Primary objective of this study is to allow access and evaluate the safety of crizotinib for patients in Japan with advanced NSCLC harboring a translocation or inversion involving the ROS1 oncogene.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of NSCLC that is locally advanced or metastatic.
* Positive for translocation or inversion events involving the ROS1 gene as determined by protocol defined test.
* ECOG performance status 0 to 2.
* Adequate organ function
* Patients with brain metastases are eligible if neurologically stable for at least 2 weeks and have no ongoing requirement for corticosteroids.
* Male patients able to father children and female patients of childbearing potential and at risk for pregnancy must agree to use 2 highly effective methods of contraception throughout the study and for at least 90 days after the last dose of crizotinib.

Exclusion Criteria:

* Currently receiving crizotinib or any investigational products.
* Prior therapy specifically directed against ROS1 fusion genes including crizotinib.
* Carcinomatous meningitis or leptomeningeal disease.
* Spinal cord compression unless treated with the patient attaining good pain control and stable or recovered neurologic function.
* Ongoing uncontrolled congestive heart failure (CHF) and any of the following within the 3 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, or cerebrovascular accident including transient ischemic attack.
* Ongoing cardiac dysrhythmias of CTCAE Grade 2, uncontrolled atrial fibrillation of any grade, or QTc more than 480 msec.
* History of extensive disseminated/bilateral or known presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not history of prior radiation pneumonitis.
* Pregnant female patients; breastfeeding female patients.
* Use of drugs or foods including known potent CYP3A4 inhibitors, known potent CYP3A4 inducers and CYP3A4 substrates with narrow therapeutic indices

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hyogo Cancer Center, Akashi, Hyōgo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081064&StudyName=Crizotinib+%28xalkori+%28registered%29%29+Expanded+Access+Protocol+For+The+Treatment+Of+Japanese+Patients+With+Advanced+Non-small+Cell+Lung+Cancer+%28nsclc%29+Harboring+A+Translocation+Or+Inversion+Involving+The+Ros1+Oncogene